CLINICAL TRIAL: NCT01769443
Title: A Prospective, Randomized, Multicenter, Two-Parallel Arm Study Evaluating the Overall Efficacy and Safety of Desensitization Therapy on Selected Patients Awaiting Heart Transplantation
Brief Title: Safety and Efficacy of Desensitization Therapy in Sensitized Participants Awaiting Heart Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to enroll within funding period
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-13; U01AI063594 (NIH)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Primary Heart Transplant; Heart Transplantation; Heart Transplant
Keywords: desensitization therapy; bortezomib (VELCADE®); plasmapheresis
MeSH Terms: interventions — Bortezomib; Plasmapheresis; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Desensitization Therapy (No Intervention): Subject(s) randomized to no desensitization therapy pre-transplant.
- Desensitization Therapy (Experimental): Subject(s) randomized to desensitization therapy pre-transplant.
  Desensitization therapy regimen pre-transplant: Plasmapheresis for 3 consecutive days (treatment days 0, 1 and 2) followed by concomitant bortezomib dosed at 1.3 mg/m^2 as a 3 to 5 second bolus intravenous injection on treatment days 0, 3, 7 and 10. The first dose of bortezomib is administered between 4-8 hours after the first plasmapheresis session is completed and there must be at least 96 hours between the second and third dose of bortezomib.
  Interventions: Drug: bortezomib; Procedure: plasmapheresis

INTERVENTIONS:
Drug: bortezomib — Bortezomib dosed at 1.3 mg/m^2 as a 3 to 5 second bolus administered by intravenous injection on treatment days 0, 3, 7 and 10. The first dose of bortezomib is administered between 4-8 hours after the first plasmapheresis session is completed and there must be at least 96 hours between the second and third dose of bortezomib.
  Other Names: VELCADE®
  Arms: Desensitization Therapy
Procedure: plasmapheresis — Plasmapheresis for 3 consecutive days (treatment days 0, 1 and 2) followed by concomitant bortezomib dosed at 1.3 mg/m^2 as a 3 to 5 second bolus administered by intravenous injection on treatment days 0, 3, 7 and 10. The first dose of bortezomib is administered between 4-8 hours after the first plasmapheresis session is completed and there must be at least 96 hours between the second and third dose of bortezomib.
  Other Names: apheresis (plasma)
  Arms: Desensitization Therapy

SUMMARY:
The primary objective is to evaluate the efficacy of desensitization therapy, which includes VELCADE® (bortezomib) and plasmapheresis, on select sensitized patients awaiting heart transplantation.

DETAILED DESCRIPTION:
Bortezomib works by decreasing plasma cells in the blood. Plasma cells produce antibodies. Plasmapheresis is a procedure that removes antibodies from the blood. Plasma cells and antibodies produced by plasma cells can be involved in organ rejection after transplantation.

This trial will evaluate if decreasing plasma cells and antibodies with bortezomib and plasmapheresis can reduce complications while participants are waiting for their heart transplant. The evaluation of efficacy is defined by a lower complication rate while on the heart transplant waitlist.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to understand and provide informed consent;
* Candidate (as recipient) for a primary heart transplant (single organ transplant);
* Calculated panel reactive antibody (cPRA) of greater than 30% with a threshold using mean fluorescent intensity (MFI) of 3,000 or standard fluorescence intensity (SFI) of 60,000;
* Status 1 (1A or 1B) enrollment and randomization to occur within 2 weeks after status 1 listing;
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse;
* Male subjects, even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse;
* Negative test for HIV (human immunodeficiency virus), HBsAg (hepatitis B surface antigen), HBcAb (hepatitis B core antibody), and HCV (hepatitis C virus) antibodies within 6 months prior to study entry.

Exclusion Criteria:

* Recipient of multiple solid organ or tissue transplants;
* Prior history of organ transplantation;
* Women of childbearing potential with a positive serum β-human chorionic gonadotropin (β-hCG) pregnancy test.Pregnancy testing is not required for postmenopausal or surgically sterilized women;
* Currently breast-feeding a child or plans to become pregnant during the timeframe of the study follow-up period;
* Subject has a hypersensitivity to VELCADE® (bortezomib), boron, or mannitol;
* Active systemic infection at time of enrollment;
* Any history of serologic positivity to HIV, HBsAg, HBcAb and HCV Ab;
* History of malignancy except when noted by an oncology specialist that tumor recurrence is low based on tumor type, response to therapy and negative metastatic work-up;
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy;
* Subjects with a platelet count of less than 75,000 within 7 days prior to enrollment;
* Subjects with an absolute neutrophil count (ANC) of less than 1,500 within 7 days prior to enrollment;
* Subjects with >1.5 x ULN (upper limit of normal) total bilirubin;
* Subjects with any grade or history of neuropathy;
* Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements;
* Participation in another interventional clinical trial or requiring treatment using un-marketed investigational drug(s) within 14 days of start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon A Kobashigawa, MD, Study Chair — Cedars-Sinai Heart Institute; Peter S. Heeger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (14):
- United States (14):
  - Cedars Sinai Heart Institute, Beverly Hills, California
  - University of California at San Francisco, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] John R, Lietz K, Burke E, Ankersmit J, Mancini D, Suciu-Foca N, Edwards N, Rose E, Oz M, Itescu S. Intravenous immunoglobulin reduces anti-HLA alloreactivity and shortens waiting time to cardiac transplantation in highly sensitized left ventricular assist device recipients. Circulation. 1999 Nov 9;100(19 Suppl):II229-35. doi: 10.1161/01.cir.100.suppl_2.ii-229. PMID 10567309
- [Background] Jordan SC, Vo A, Bunnapradist S, Toyoda M, Peng A, Puliyanda D, Kamil E, Tyan D. Intravenous immune globulin treatment inhibits crossmatch positivity and allows for successful transplantation of incompatible organs in living-donor and cadaver recipients. Transplantation. 2003 Aug 27;76(4):631-6. doi: 10.1097/01.TP.0000080685.31697.FC. PMID 12973100
- [Background] Leech SH, Lopez-Cepero M, LeFor WM, DiChiara L, Weston M, Furukawa S, Macha M, Singhal A, Wald JW, Nikolaidis LA, McClurken JB, Bove AA. Management of the sensitized cardiac recipient: the use of plasmapheresis and intravenous immunoglobulin. Clin Transplant. 2006 Jul-Aug;20(4):476-84. doi: 10.1111/j.1399-0012.2006.00509.x. PMID 16842525
- [Background] McGee EC Jr, Cotts W, Tambur AR, Friedewald J, Kim J, O'Connell J, Wallace S, McCarthy PM. Successful bridge to transplant in a highly sensitized patient with a complicated pump pocket infection. J Heart Lung Transplant. 2008 May;27(5):568-71. doi: 10.1016/j.healun.2008.02.006. PMID 18442726
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/Pages/default.aspx
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study planned to enroll 80 participants; however, the decision to terminate the study was made due to the very slow rate of participant accrual and the inability to meet the recruitment goal within the funding period. Only 2 participants were enrolled at one site before study recruitment status changed to "Active, not recruiting."
Groups:
- No Desensitization: No desensitization therapy pre-transplantation
- Desensitization: Plasmapheresis with concomitant bortezomib.
  * Plasmapheresis will be given for 3 consecutive days (treatment days 0, 1 and 2) within 2 weeks of Status I listing for heart transplantation. Plasmapheresis is a procedure that involves the extracorporeal separation of plasma from cellular blood components by centrifugation or membrane filtration, which removes the alloantibody. The plasma depleted blood is reconstituted with exogenous fresh-frozen plasma or albumin solution which is then infused back into the patient.
  * Four doses of bortezomib (1.3 mg/m^2) were administered intravenously on treatment days 0, 3, 7 and 10. The first dose was given between 4-8 hours after the first plasmapheresis session was completed and there was at least 96 hours between the second and third dose of bortezomib
Period: Overall Study
Arm/Group | No Desensitization | Desensitization
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Study closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | No Desensitization | Desensitization | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Composite of Incidence of the Following Events in Subjects
Description: * Death,
  * Removal from the transplant waiting list for any reason except improvement of cardiac function,
  * Initiation of any mechanical circulatory support device,
  * Severe infection requiring intravenous antibiotics,
  * Cerebral vascular accident,
  * Acute renal failure requiring dialysis.
Time Frame: At transplant, or 90 days post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time From Wait Listing to Heart Transplantation
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Calculated PRA (cPRA) From Wait Listing to Transplantation
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Death
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Removal From Transplant Waiting List for Any Reason Except Improvement of Cardiac Function
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Initiation of Any Mechanical Circulatory Support Device
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Severe Infection Requiring Intravenous Antibiotics
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Incidence of Cerebral Vascular Accident
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Incidence of Acute Renal Failure Requiring Hemodialysis
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence of Administering Desensitization Therapy Beyond 90 Days After Randomization
Time Frame: At transplant, or 1 year post-randomization, whichever occurs first
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Development of Angiographically Evident Cardiac Allograft Vasculopathy at 1 Year
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Incidence of Serious Infections Requiring Intravenous Antimicrobial Therapy
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Subjects on Left Ventricular Assist Devices (LVAD) Compared to Those Not on LVADs
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Cardiac Dysfunction as Reflected in the Left Ventricular Ejection Fractions < 40% by Echocardiography, Angiogram or Nuclear Testing.
Time Frame: 24 and 52 weeks:
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Incidence of Post-Transplant Lymphoproliferative Disorder (PTLD)
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Death
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Re-transplantation or Re-listed for Transplantation
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Groups:
- Desensitization: Plasmapheresis with concomitant bortezomib.
  * Plasmapheresis will be given for 3 consecutive days (treatment days 0, 1 and 2) within 2 weeks of Status I listing for heart transplantation. Plasmapheresis is a procedure that involves the extracorporeal separation of plasma from cellular blood components by centrifugation or membrane filtration, which removes the alloantibody. The plasma depleted blood is reconstituted with exogenous fresh-frozen plasma or albumin solution which is then infused back into the patient.
  * Four doses of bortezomib (1.3 mg/m2) were administered intravenously on treatment days 0, 3, 7 and 10. The first dose was given between 4-8 hours after the first plasmapheresis session was completed and there was at least 96 hours between the second and third dose of bortezomib
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Incidence of Hospitalizations
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Incidence of Rejection Episodes Per Subject and Freedom From Rejection
Description: Rejection is defined as follows:
  * Biopsy proven acute rejection (BPAR) of any grade (cellular rejection per 2004 ISHLT [International Society of Heart and Lung Transplantation] grading scale),
  * BPAR (individual grades),
  * BPAR (Biopsy Proven Acute Rejection) > 2R
  * antibody mediated rejection (AMR),
  * Any treated rejection,
  * Rejection associated with hemodynamic compromise (HDC).
Time Frame: 24 and 52 weeks post-transplantation
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | No Desensitization | Desensitization
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the first protocol mandated procedure until the study completion, or until 30 days after the subject prematurely withdraws from the study.
Description: The participant randomized to the control arm ("No Desensitization Therapy") completed week 24 (6 months) of post-transplantation evaluations. The participant assigned to the Investigational Arm ("Desensitization Therapy") completed week 52 (12 months) of post-transplantation follow-up.
Arm/Group | No Desensitization | Desensitization
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Desensitization (N=1) | Desensitization (N=1)
compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated by the study sponsor, with agreement from the investigators. Reason: very slow rate of accrual and inability to meet the accrual goal within the funding period. (N=2 enrolled. Aim was 80 participants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No